CLINICAL TRIAL: NCT03052530
Title: Sapphire II PRO - A Prospective, Open Label, Multi-center, Single Arm, Observational Study Designed to Evaluate the Acute Safety and Device Procedural Success of the Sapphire II PRO 1.0 and 1.25 mm PTCA Dilatation Catheters.
Brief Title: Sapphire II PRO US Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrbusNeich (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-0714
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Results first posted 2018-04-04 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sapphire II PRO (Experimental): Single arm with investigational Sapphire II PRO 1.0 and 1.25 mm PTCA dilatation catheters
  Interventions: Device: Sapphire II PRO

INTERVENTIONS:
Device: Sapphire II PRO — To pre-dilate coronary arteries or bypass grafts during the subject's index procedure with Sapphire II PRO 1.0 and 1.25 PTCA dilatation catheters.

SUMMARY:
A prospective, open label, multi-center, single arm, observational study designed to evaluate the acute safety and device procedural success of the Sapphire II PRO 1.0 and 1.25 mm PTCA dilatation catheters in subjects with stenotic coronary arteries or bypass grafts during percutaneous coronary intervention.

Sixty (60) subjects will be treated at up to 5 U.S. sites with the Sapphire II PRO diameters 1.0 and 1.25 mm PTCA dilatation catheters to pre-dilate coronary arteries or bypass grafts during their index procedure. All subjects will be screened according to the protocol inclusion and exclusion criteria and will be followed through hospital discharge.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedures.
3. Subject must agree not to participate in any other clinical study during hospitalization for the index procedure that would interfere with the endpoints of this study.
4. Subjects must have a single or double vessel coronary artery disease and clinical evidence of ischemic heart disease, such as stable / unstable angina or silent ischemia.

   Angiographic Inclusion Criteria
5. Subject must have de novo or restenotic lesion(s) in native coronary arteries or bypass grafts that are suitable for percutaneous coronary intervention. An embolic protection device must be used in all Saphenous venous grafts (SVG) interventions performed during the index procedure.
6. A maximum of two lesions, including at least one target lesion, in up to two coronary arteries.
7. Target and non-target lesions must be located in different coronary arteries or bypass grafts.
8. Target lesion(s) must have a diameter stenosis of ≥70% by visual estimation and may include chronic total occlusions (CTO)
9. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success.

Clinical Exclusion Criteria:

1. Subject with a known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, anti-platelet medications, or sensitivity to contrast media which cannot be adequately pre-medicated.
2. Subject with known diagnosis of an acute myocardial infarction (AMI) within 72 hours prior to index procedure.
3. Subject with known pregnancy or is nursing. Women of child- bearing potential should have a documented negative pregnancy test within 7 days before index procedure.
4. Planned or actual target lesion treatment with an unapproved device, atherectomy, laser, cutting balloon or thrombectomy during the index procedure.
5. A serum creatinine level > 2.0 mg/dl within seven days prior to index procedure.
6. Cerebrovascular accident (CVA) within the past 6 months.
7. Active peptic ulcer or active gastrointestinal (GI) bleeding within the past 6 months.
8. Subject has a known left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown, if necessary)

   Angiographic Exclusion Criteria
9. More than two lesions requiring treatment.
10. Unprotected left main coronary artery disease.(Greater than 50% diameter stenosis)
11. Coronary artery spasm of the target vessel in the absence of a significant stenosis.
12. Target lesion with angiographic presence of probable or definite thrombus.
13. Target lesion involves a bifurcation requiring treatment with more than one stent or pre-dilatation of a side branch >2.0 mm in diameter.
14. Non-target lesion to be treated during the index procedure meets any of the following criteria:

    * Located within a bypass graft (venous or arterial)
    * Left main location
    * Chronic total occlusion
    * Involves a bifurcation (e.g., bifurcations requiring treatment with more than 1 stent)
    * Treatment not deemed a clinical angiographic success

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (4):
- United States (4):
  - University of Miami, Miami, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - The Christ Hospital Heart and Vascular, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sapphire II PRO
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sapphire II PRO
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.26 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 3
  White | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61
Cardiac History [Count of Participants; unit: Participants] — More than one Cardiac History measure may be reported for each participant.
  Participants
    Previous Percutaneous Coronary Intervention | 31
    Previous Coronary Artery Bypass Graft | 18
    Previous Myocardial Infarction | 25
    Stable Angina | 31
    Unstable Angina | 21
Cardiac Risk Factors [Count of Participants; unit: Participants] — More than one Cardiac Risk Factor may be reported for each participant.
  Participants
    Current Cigarette Smoking (within 30 days) | 10
    Medically Treated Diabetes | 16
    Hypercholesterolemia Requiring Treatment | 55
    Hypertension Requiring Treatment | 51
Lesion Characteristics: Vessel Treated [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    Bypass Graft | 4
    Diagonol Branch-Left Anterior Descending Artery | 10
    Left Anterior Descending Artery | 22
    Left Circumflex Artery | 12
    Marginal Branch of Left Circumflex Artery | 1
    Posterior Descending Branch-Right Coronary Artery | 2
    Right Coronary Artery | 16
Lesion Characteristics: Lesion Location [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    Distal | 11
    Mid | 27
    Ostial | 3
    Prox | 26
Lesion Characteristics [Mean (Standard Deviation); unit: Millimeters] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Millimeters
    Lesion Length | 18.42 (12.25)
    Minimum Lumen Diameter | .52 (.35)
Lesion Characteristics [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    Thrombus | 1
    Tortuosity | 0
    Calcification | 34
    Ulceration | 4
    Aneurysm | 0
    Total Occlusion | 9
Lesion Characteristics: Pre-Procedure Thrombolysis in Myocardial Infarction (TIMI) Flow [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    0 (no perfusion) | 9
    1 (penetration with minimal perfusion) | 4
    2 (partial perfusion) | 4
    3 (complete perfusion) | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device Procedural Success
Description: Device procedural success consisting of the following:
  * Successful delivery, inflation, deflation and withdrawal of the study balloon
  * No evidence of vessel perforation, flow limiting dissection (grade C or higher) or reduction in TIMI flow from baseline related to the study balloon
  * Final TIMI flow grade of 3 at the conclusion of the PCI procedure
Time Frame: Peri-procedural (at Day 0)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapphire II PRO
Number analyzed (Participants) | 61
Participants | 59

2. Secondary Outcome: Number of Participants With In-hospital Major Adverse Cardiac Events (MACE)
Description: In-hospital Major Adverse Cardiac Events (MACE)
  * All death (cardiac and non-cardiac)
  * Myocardial infarction (MI)
  * Target Lesion Revascularization (TLR)
Time Frame: Endpoints will be measured through hospital discharge (expected to be within 24 hours)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapphire II PRO
Number analyzed (Participants) | 61
Participants | 1

3. Secondary Outcome: Number of Participants With In-hospital Stent Thrombosis (ST) Within the Target Vessel
Description: In-hospital stent thrombosis (ST) within the target vessel
Time Frame: Endpoint will be measured through hospital discharge (expected to be within 24 hours)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapphire II PRO
Number analyzed (Participants) | 61
Participants | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Arrhythmias (Requiring Intervention)
Description: Clinically Significant Arrhythmias (requiring intervention)
Time Frame: Endpoint will be measured through hospital discharge (expected to be within 24 hours)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapphire II PRO
Number analyzed (Participants) | 61
Participants | 0

ADVERSE EVENTS:
Time Frame: Per the protocol, adverse events were collected from the point of subject enrollment through study completion at hospital discharge (hospital stay expected to be an average of 24 hours).
Arm/Group | Sapphire II PRO
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 1/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sapphire II PRO (N=61)
Myocardial infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03052530/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03052530/SAP_001.pdf